CLINICAL TRIAL: NCT06938919
Title: Impact of Implementing an Electronic Respiratory Sound Monitoring System for Quality Improvement in Gastrointestinal Endoscopic Sedation: A Randomized Controlled Trial
Brief Title: Electronic Respiratory Sound Monitoring System in Gastrointestinal Endoscopic Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Metal Industries Research & Development Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202409073DINC
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-04

CONDITIONS: Gastrointestinal Endoscope; Endoscopic Retrograde Cholangiopancreatogram (ERCP)
Keywords: Electronic repiratory sound monitoring system; Gstrointestinal endoscopic sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): routine care
  Interventions: Device: routine care without electronic respiratory sound monitoring system
- Experimental (Experimental): routine care combine with electronic respiratory sound monitoring system
  Interventions: Device: routine care with electronic respiratory sound monitoring system

INTERVENTIONS:
Device: routine care without electronic respiratory sound monitoring system — Maintain heart rate between 50-100 bpm; maintain systolic blood pressure between 90-160 mmHg; maintain SpO2 above 94%.
  Arms: Control group
Device: routine care with electronic respiratory sound monitoring system — Maintain heart rate between 50-100 bpm; maintain systolic blood pressure between 90-160 mmHg; maintain SpO2 above 94%; and refer to the following electronic breath sound abnormalities to maintain sedation depth: Maintain respiratory rate (RR) at 12-20 bpm; avoid partial airway obstruction
  Arms: Experimental

SUMMARY:
This study aims to evaluate the application of an electronic respiratory sound monitoring system during sedation for gastrointestinal endoscopy and to determine its effectiveness in improving sedation quality. Gastrointestinal endoscopy is a common medical procedure, but respiratory complications caused by sedation, such as hypoventilation and airway obstruction, are significant safety concerns. Traditional respiratory monitoring methods, such as end-tidal CO2 monitoring, are often unreliable due to difficulties in gas sampling during the procedure. In contrast, an electronic respiratory sound monitoring system can accurately capture tracheal breathing sounds and provide important parameters such as respiratory rate and airway obstruction ratio, helping clinicians avoid over-sedation. This study will conduct a randomized controlled trial with 120 participants, divided into a control group with conventional monitoring and an experimental group using the electronic respiratory sound monitoring system. The study will compare sedation dosage, airway complications, and recovery speed between the two groups, and further analyze the clinical value of the system's parameters. The findings of this study will contribute to improving the safety and precision of sedation during gastrointestinal endoscopy and provide evidence for future clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo routine colonoscopy plus gastroscopy or endoscopic retrograde cholangiopancreatography (ERCP) and require deep sedation

Exclusion Criteria:

* Pregnancy
* Patients diagnosed with sleep apnea or morbid obesity (BMI greater than 40 kg/m2)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Desaturation | during the procedure
  Incidence and duration of SpO2< 94%

SECONDARY OUTCOMES:
Incidence of airway management for desaturation | during the procedure
  jaw thrust manuever, nasal airway insertion, mask ventilation
Total amount of anesthetics | during the procedure
  Total amount of anesthetics used

OTHER OUTCOMES:
QoR-15 Questionnaire | 24 hours
  QoR-15 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Cheng Chan, M.D.,PhD., Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No